CLINICAL TRIAL: NCT02205034
Title: Evaluation of Tolerance, Suckling and Food Intake After Repeated Nasals Administrations of Oxytocin in PWS Infants
Acronym: OTBB2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12 391 02; 1239102 (Other Grant/Funding Number: Toulouse University Hospital Funding)
Record Dates: First submitted 2014-07-22; First posted 2014-07-31 (Estimated); Results first posted 2023-12-04 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-01

CONDITIONS: Prader Willi Syndrome
Keywords: Prader Willi
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- first arm (Active Comparator): 4IU of oxytocin every other day
  Interventions: Drug: oxytocin
- second arm (Active Comparator): 4 IU of oxytocin daily
  Interventions: Drug: oxytocin
- third arm (Active Comparator): 4 IU of oxytocin twice daily
  Interventions: Drug: oxytocin

INTERVENTIONS:
Drug: oxytocin — Intranasal administration
  Other Names: Oxytocin (Syntocinon)

SUMMARY:
The Prader-Willi syndrome (PWS) includes severe neonatal hypotonia with impaired suckling leading to failure to thrive in the most severe cases, subsequently followed by an early onset of morbid obesity with hyperphagia and deficit of satiety, combined with other endocrine dysfunction probably due to hypothalamic dysfunction. The pathophysiological mechanism of the occurrence of the 2 main nutritional phases of PWS is unknown. Swaab reported a deficit in the oxytocin (OT)-producing neurons of the paraventricular nucleus in the brain of these patients. In addition of its well-known anorexigenic effect, OT is involved in establishing and maintaining social codes. Moreover in a PWS mouse model generated from a MAGEL2 KO gene a single OT injection at 5 hr of life prevent the early death observed in 50 % of the new born mice by recovering normal suckling. Interestingly this effect is no longer observed if OT injection takes place later. Our hypothesis is that early administration of OT in babies with PWS may improve suckling and possibly infant-mother interactions. In our recent study (manuscript in preparation), we have shown that a single intranasal administration of OT is well tolerated. This escalating dose study is designed to evaluate the tolerance of repeated intranasal administration of OT in 3 steps (4IU every other day, 4 IU daily, 4IU twice daily) in babies younger than 5 months with PWS.

DETAILED DESCRIPTION:
Prader-Willi syndrome (PWS) is a rare, complex multisystem genetic disorder arising from the lack of expression of paternally inherited imprinted genes on chromosome 15q11-q13. The syndrome includes severe neonatal hypotonia with impaired suckling leading to failure to thrive in the most severe cases, subsequently followed by an early onset of morbid obesity with hyperphagia and deficit of satiety, combined with other endocrine dysfunction probably due to hypothalamic dysfunction. The pathophysiological mechanism of the occurrence of the 2 main nutritional phases of PWS is unknown. Swaab reported a deficit in the oxytocin (OT)-producing neurons of the paraventricular nucleus in the brain of these patients. In addition of its well-known anorexigenic effect, OT is involved in establishing and maintaining social codes. Moreover in a PWS mouse model generated from a MAGEL2 KO gene a single OT injection at 5 hr of life prevent the early death observed in 50 % of the new born mice by recovering normal suckling. Interestingly this effect is no longer observed if OT injection takes place later. Our hypothesis is that early administration of OT in babies with PWS may improve suckling and possibly infant-mother interactions. In our recent study (manuscript in preparation), we have shown that a single intranasal administration of OT is well tolerated. This escalating dose study is designed to evaluate the tolerance of repeated intranasal administration of OT in 3 steps (4IU every other day, 4 IU daily, 4IU twice daily) in babies younger than 5 months with PWS.

ELIGIBILITY:
Inclusion Criteria:

* Infants with PWS genetically confirmed
* Aged less than 5 months

Exclusion Criteria:

* Infants presenting hepatic insufficiency
* Infants presenting renal insufficiency
* Infants with abnormal ECG

Ages: 1 Month to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maïthé TAUBER, Principal Investigator — Endocrinologie pédiatrique, Hospital of Toulouse
Locations (1):
- Centre de réfrence Prader-Willi, Hospital of infants, Toulouse, France

REFERENCES:
- [Result] Tauber M, Boulanouar K, Diene G, Cabal-Berthoumieu S, Ehlinger V, Fichaux-Bourin P, Molinas C, Faye S, Valette M, Pourrinet J, Cessans C, Viaux-Sauvelon S, Bascoul C, Guedeney A, Delhanty P, Geenen V, Martens H, Muscatelli F, Cohen D, Consoli A, Payoux P, Arnaud C, Salles JP. The Use of Oxytocin to Improve Feeding and Social Skills in Infants With Prader-Willi Syndrome. Pediatrics. 2017 Feb;139(2):e20162976. doi: 10.1542/peds.2016-2976. PMID 28100688
- [Result] Viaux-Savelon S, Rosenblum O, Guedeney A, Diene G, Cabal-Berthoumieu S, Fichaux-Bourin P, Molinas C, Faye S, Valette M, Bascoul C, Cohen D, Tauber M. Dyssynchrony and perinatal psychopathology impact of child disease on parents-child interactions, the paradigm of Prader Willi syndrom. J Physiol Paris. 2016 Nov;110(4 Pt B):427-433. doi: 10.1016/j.jphysparis.2017.08.001. Epub 2017 Sep 1. PMID 28823614
- [Derived] Borie AM, Dromard Y, Guillon G, Olma A, Manning M, Muscatelli F, Desarmenien MG, Jeanneteau F. Correction of vasopressin deficit in the lateral septum ameliorates social deficits of mouse autism model. J Clin Invest. 2021 Jan 19;131(2):e144450. doi: 10.1172/JCI144450. PMID 33232306

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | First Arm | Second Arm | Third Arm
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First Arm | Second Arm | Third Arm | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 6 | 18
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4 | 8
  Male | 3 | 5 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Occurence of Adverse Event
Description: Occurrence of adverse event, description and quantification of their severity, imputability to repeated intranasal administration of OT (4IU every other day, 4 IU daily, 4IU twice daily) during the 7 days following the first administration.
Time Frame: up to day 8 (Visit 8)
Measure: Number; unit: number of adverse events
Arm/Group | First Arm | Second Arm | Third Arm
Number analyzed (Participants) | 6 | 6 | 6
number of adverse events | 10 | 9 | 6

2. Secondary Outcome: NOMAS Score
Description: NOMAS score evaluate sucking/swallowing abilitites of infants during feeding; endpoint is the % of infants who reached a NOMAS score <= 10 (normal score)
Time Frame: Before and after 7 days of treatment
Reporting Status: Not Posted

3. Secondary Outcome: Videofluoroscopy of Swallowing Score
Description: Videofluoroscopy of swallowing score (VFSS score)
Time Frame: before and after 7 days of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: everyday during the trial so during 7 days
Arm/Group | First Arm | Second Arm | Third Arm
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 5/6 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Arm (N=6) | Second Arm (N=6) | Third Arm (N=6)
Pneumopathy (Infections and infestations) | 1 (1) | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Arm (N=6) | Second Arm (N=6) | Third Arm (N=6)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastro-oesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Culture urine positive (Investigations) | 0 (0) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Oral candidasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infantile colic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes